CLINICAL TRIAL: NCT03355092
Title: vBloc Therapy for Obese Subjects With Type 2 Diabetes- A Randomized Controlled Clinical Trial
Brief Title: The vBlocT2D Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPSC IRB 11343; KPSC IRB 11343 (Other: Kaiser Permanente Southern California IRB)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Type2 Diabetes; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- vBloc Therapy + Usual Care for Type 2 Diabetes (Experimental)
  Interventions: Device: vBloc Therapy
- Usual Care for Type 2 Diabetes (No Intervention)

INTERVENTIONS:
Device: vBloc Therapy — The vBloc device will be placed using a laparoscopic procedure. The participants will be followed according to standard clinical practice and vBloc therapy protocol under the supervision of study surgeons. . Pre-operative testing will be conducted per surgeon's evaluation. Participants will receive weight management education according to the vBloc Therapy protocol.
  Arms: vBloc Therapy + Usual Care for Type 2 Diabetes

SUMMARY:
Overall aim: To demonstrate that weight loss through vBloc Therapy in combination with usual care will achieve better glycemic control for patients with obesity and type 2 diabetes than usual care alone.

Duration: Participants will be asked to participate in a 12 month study that involves a baseline visit and research follow-up visits at 3, 6, 9, and 12 months.

Sample Size: 60 participants will be enrolled in the study. Of these, 30 will be randomized to vBloc therapy and 30 will be randomized to usual care.

DETAILED DESCRIPTION:
The vBlocT2D study is a two arm, randomized, controlled, unblinded clinical trial in which 60 adult patients with T2D with moderate to extreme obesity (BMI 35-45 kg/m2) and suboptimal glycemic control (glycated haemoglobin (HbA1c) 7-10%) without significant diabetic complications, will be randomized to usual care alone (n=30) or vBloc therapy plus usual care (n=30) to assess the superiority of vBloc therapy plus usual care than standard usual care alone in improving diabetic control. The vBloc therapy will be delivered through an electrical and reversible vagal blocking device (the Maestro Rechargeable System) implanted using laparoscopic surgery. The device was approved by the FDA in 2015 for weight loss in adults with BMI 40-45 kg/m2, or BMI 35-39.9 kg/m2 with one or more obesity-related co-morbid conditions. The study will recruit patients over a 12-month period and follow each individual for 12-months post intervention. The primary outcome is change in HbA1c at 12-months post randomization. The secondary outcomes are changes in weight, waist and hip circumferences, blood pressure, lipids, insulin sensitivity and β-cell health measured through oral glucose tolerance testing, dietary intake, eating behaviors, physical activity, quality of life and potential circulating biomarkers. Medication use, clinical labs and adverse events will be compared as well.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes with HbA1c level 7-10% inclusive, AND known duration of disease ≤10 years, AND
2. Male or female (females of child-birth potential not pregnant at implant or for duration of study), AND
3. Age 18 years or older, AND
4. Body mass index (BMI) 35-45 kg/m2 inclusive, AND
5. Attempt and failed diet, exercise and behavioral modification program within past five years,

Exclusion Criteria:

1. Use of GLP-1 receptor agonists for diabetes currently or within past 6 months
2. Contraindications to vBloc (permanently implanted, electrical-powered medical device or gastrointestinal device or prosthesis (e.g. pacemakers, implanted defibrillators, neurostimulators))
3. Patients for whom magnetic resonance imaging (MRI), shortwave, microwave, or therapeutic ultrasound diathermy is planned (Note: Diathermy is any treatment that uses high-frequency electromagnetic radiation, electric currents, or ultrasonic waves to produce heat in body tissues. Patients absolutely CANNOT be treated with any type of shortwave, microwave, or therapeutic ultrasound diathermy device whether or not it is used to produce heat. These treatments should not be applied anywhere on the body)
4. Underlying disease(s) likely to (a) limit life span to less than study duration and/or (b) increase risk of intervention outside of the study and/or (c) limit ability to participate in outcomes assessment and/or (d) limit participation
5. Previous bariatric or upper GI surgery
6. Excessive alcohol intake
7. Current smokers or smoking cessation in prior 3 months
8. An underlying disease known to have important effects on glucose metabolism
9. Active infections
10. Anemia (Hemoglobin <11g/dl in women, <12 g/dl in men) or known coagulopathy
11. Chronic kidney disease manifest as serum creatinine >2.0 mg/dl
12. Diabetic retinopathy requiring photocoagulation therapy
13. Symptomatic diabetic gastroparesis
14. Cardiovascular disease, including uncontrolled hypertension and symptomatic congestive heart failure
15. Cirrhosis of the liver, portal hypertension, or esophageal varices
16. Symptomatic esophageal reflux
17. Conditions or behaviors likely to affect the conduct of the vBloc Study

    1. Unable or unwilling to give informed consent
    2. Unable to adequately communicate with clinic staff
    3. Current or anticipated participation in another intervention research project that would interfere with any of the interventions/outcomes in vBloc study
    4. Likely to move away from participating clinic in next 2 years
    5. Current (or anticipated) pregnancy and lactation.
    6. Major psychiatric disorder that, in the opinion of investigators, would impede participation in the study
    7. Weight loss >7% in past two months for any reason except postpartum weight loss.
18. Additional conditions may serve as criteria for exclusion at the discretion of the study investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Mean reduction in HbA1c | at 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anny Xiang, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente South Bay Medical Center, Harbor City, California, United States